CLINICAL TRIAL: NCT07010497
Title: A PHASE 2, OPEN-LABEL STUDY OF IRPAGRATINIB IN COMBINATION WITH ATEZOLIZUMAB AND BEVACIZUMAB IN PATIENTS WITH ADVANCED OR UNRESECTABLE HEPATOCELLULAR CARCINOMA (IAPETUS)
Brief Title: A Prospective Study to Evaluate the Safety and Efficacy of the Combination Therapy of Irpagratinib, Atezolizumab, and Bevacizumab in Patients With Hepatocellular Carcinoma
Acronym: IAPETUS
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Asan Medical Center (Other)
Collaborators: Abbisko Therapeutics Co, Ltd (Industry)
Responsible Party: Principal Investigator, Changhoon Yoo, Associate Professor, Asan Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ABSK-011-2001
Record Dates: First submitted 2025-05-15; First posted 2025-06-08 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-05

CONDITIONS: Carcinoma, Hepatocellular
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- irpagratinib (Experimental): Atezolizumab: 1200 mg on Day 1 of each 21-day cycle. Bevacizumab: 15 mg/kg on Day 1 of each 21-day cycle. ABSK-011 (irpagratinib): Patients will receive oral administration of ABSK-011 in a repetitive dosing regimen for a period of 21 consecutive days as a cycle, either once daily or twice daily, until the investigators make a comprehensive assessment of imaging examinations, laboratory data, and the clinical condition of the patients, and determine that there is intolerable toxicity or disease progression.
  Interventions: Drug: irpagratinib

INTERVENTIONS:
Drug: irpagratinib — Patients will receive oral administration of ABSK-011 capsules in a repetitive dosing regimen for a period of 21 consecutive days as a cycle, either once daily or twice daily, until the investigators make a comprehensive assessment of imaging examinations, laboratory data, and the clinical condition of the patients, and determine that there is intolerable toxicity or disease progression.

SUMMARY:
This is a phase 2, open-label study to evaluate the safety, tolerability and efficacy of Irpagratinib in combination with Atezolizumab and Bevacizumab in patients with advanced or unresectable HCC harboring FGF19 overexpression.

This study composes two parts, a Safety Run-in part to evaluate safety and establish the dose of Irpagratinib for the triple combination, and an Expansion part to evaluate the preliminary efficacy and safety using Simon's two-stage design.

DETAILED DESCRIPTION:
Safety Run-in This part will enroll 9 patients administered with Irpagratinib orally 150 mg BID or 200 mg BID from study ABSK-011-101 in repeated 21-day cycles, plus Atezolizumab 1200 mg and Bevacizumab 15 mg/kg given IV Q3W. The tolerability will be evaluated upon the incidence of DLTs observed during Cycle 1. If DLT happened in ≤1 of the 3 DLT evaluable patients in 150 mg BID cohort, a combination regimen cohort with Irpagratinib orally 200 mg BID plus Atezolizumab 1200 mg Q3W+ Bevacizumab 15mg/kg Q3W will be initiated in additional 6 DLT evaluable patients to observe the incidence of DLTs. If DLT happened in ≤1 of the 6 patients in 200 mg BID, Irpagratinib 200 mg BID + Atezolizumab 1200 mg/Q3W + Bevacizumab 15mg/kg Q3W combination regimen will be recommended for the Expansion part. If DLT happened in ≥2 of the 6 DLT evaluable patients in 200 mg BID cohort and ≤1 of the 3 DLT evaluable patients in 150 mg BID, Irpagratinib 150 mg BID + Atezolizumab 1200 mg/Q3W + Bevacizumab 15mg/kg Q3W combination regimen will be recommended for the Expansion part.

Subsequent patients of Safety Run-in should be dosed at least 7 days after the first patient's (sentinel patient) first dosing for each dose level of Irpagratinib. Eventually, the dose of Irpagratinib selected for the Expansion will be confirmed safe by at least 6 DLT evaluable patients in which ≤1 DLT event happen in 200 mg BID or at least 3 DLT evaluable patients in which ≤1 DLT event happen in 150 mg BID. Adverse events that meet the DLT definition occurring beyond the DLT observation period in patients will not be taken as a DLT but will be considered as a reference for the assessment of overall safety.

Expansion Up to 24 eligible patients will be treated with Irpagratinib (the recommended dose from Safety Run-in) + Atezolizumab 1200 mg IV Q3W (dosed in 3-week cycles) and Bevacizumab 15 mg/kg IV Q3W (dosed in 3-week cycles).

The decision for running stage two of the enrollment will be made after 3 responders observed in first evaluable 9 patients with FGF19 overexpression.

Patients who interrupt or discontinue study treatments may continue the remaining treatment if the patients are experiencing clinical benefit in the opinion of the investigator and after consultation with the Investigator (e.g., patients who transiently withhold or permanently discontinue from treatment with one of the three drugs due to adverse events may continue with the remaining drug(s)).

ELIGIBILITY:
Inclusion Criteria:

* 1.Patient should understand, sign, and date the written voluntary informed consent form prior to any protocol-specific procedures performed. Patient should be able and willing to comply with study visits and procedures as per protocol.
* 2.Male or female, aged ≥19 at the time of signing inform consent form.
* 3.Patients must have histological or cytological confirmed advanced or unresectable HCC not amenable to curative surgical or loco-regional therapies. And patients must satisfy:

  1. Provide archived tissue sample for FGF19 overexpression detection.For Safety-Run in and Expansion: the result of FGF19 overexpression lab testing must be positive as defined. Only tissue from primary lesion of liver is eligible.
  2. Barcelona Clinic Liver Cancer (BCLC) stage B or C and Child-Pugh score 5~6 without hepatic encephalopathy, no clinically apparent ascites or require medical intervention.
  3. Have at least 1 target lesion (per RECIST v1.1). Patients who received prior local therapy (e.g., radiofrequency ablation, percutaneous injection, cryoablation, high-intensity focused ultrasound, transarterial (chemo) embolization, etc.) are eligible provided the target lesion(s) have not been previously treated with local therapy or the target lesion(s) within the field of local therapy have subsequently progressed per RECIST v1.1.
* 4.ECOG performance status score 0-1
* 5.Life expectancy ≥ 3 months
* 6.Adequate organ and hematologic function as indicated by the following screening assessments performed within 14 days prior to the first administration (without blood transfusion, or medication with stimulation factors or thrombopoietin receptor agonists (TPO-RAs) within 14 days before blood sample collection):a) Absolute neutrophil count (ANC) ≥1.0×109/Lb) Platelet count (PLT) ≥75×109/Lc) Hemoglobin (Hb) ≥85g/L (8.5g/dL)d) Total bilirubin (TBIL) ≤3×ULNe) Aspartate transaminase (AST) and alanine transaminase (ALT) ≤ 5 ×ULNf) Serum creatinine (Cr) ≤1.5×ULN or creatinine clearance (Crcl) ≥50 mL/min based on Cockcroft-Gault formulag) For patients not receiving therapeutic anticoagulation: International Normalized Ratio (INR) and Activated Partial Thromboplastin Time (APTT) ≤2×ULN.h) Urinalysis for proteinuria <2+ (patients discovered to have ≥2+ proteinuria on urinalysis at baseline should undergo a 24-hour urine collection and must demonstrate <1g of protein in 24 hours)
* 7.Non-surgically sterilized male or female patients of childbearing potential must agree to use effective methods of birth control during the study and for up to 6 months after the last dose of study drug. Non-surgically sterilized female patients of childbearing potential must in non-lactation period and have a negative β-HCG test result within 14 days before first administration.

Exclusion Criteria:

Prior/Concomitant Therapy

* 1. Has received any systemic chemotherapy, including anti-VEGF therapy, or any systemic investigational anticancer agents for advanced/unresectable HCC. Patient who has received one cycle of Atezolizumab plus Bevacizumab is eligible for this trial.
* 2. Has received prior therapy with immune checkpoint inhibitors or immune stimulatory agents (eg, anti-PD-1, anti-PD-L1/2, anti-CTLA-4, anti-TIGIT, OX-40, or CD137). Patients has received one cycle of Atezolizumab plus Bevacizumab is eligible for this trial.
* 3. Previous treatment with FGFR inhibitors including selective FGFR4 or pan-FGFR inhibitors.
* 4. Has received locoregional therapy to liver (transcatheter chemoembolization, transcatheter embolization, hepatic arterial infusion, radiation, radioembolization, or ablation) within 4 weeks prior to the first dose of study intervention.
* 5. Previous anti-cancer therapy prior to initiation of study treatment: major surgery (except palliative therapy), radiotherapy (bone-marrow exposure >30%), loco-regional treatment <4 weeks; endocrine therapy with anti-tumor indications for < 2 weeks.
* 6. Prior toxicities from radiotherapy and other anti-cancer therapies that have not recovered to Grade ≤1 (CTCAE v5.0) except for which eligibility criteria allowed, alopecia, vitiligo, hormone replacement therapy controlled stable hypothyroidism, and Grade ≤2 neurotoxicity or toxicities related to prior one cycle of Atezolizumab plus Bevacizumab that investigator believes don't affect patients and safety assessment.
* 7. Concomitant use of inhibitors or inducers of P-gp transporter; or strong inhibitors or inducers of CYP3A4 (including grapefruit juice, grapefruit hybrids, pomegranates, starfruits, pomelos, Seville oranges or juice or products) within at least 14 days prior to the first dose of the study drug.
* 8. Treatment with systemic corticosteroids or other systemic immunosuppressive medications (including but not limited to prednisone, dexamethasone, cyclophosphamide, azathioprine, methotrexate, thalidomide, and anti-tumor necrosis factor agents) within 2 weeks prior to initiation of study treatment, or anticipated requirement for systemic immunosuppressive medications during the trial (except for patients who received one-time, acute, low-dose prednisone <7.5 mg/d or equivalent corticosteroids).
* 9. Vaccination with a live, attenuated vaccine within 4 weeks of the first dose of study treatment and while on trial is prohibited except for administration of inactivate vaccines (e.g., COVID-19 vaccines, inactivated influenza vaccines).
* 10. Chronic daily treatment with a nonsteroidal anti-inflammatory drug (NSAID). Occasional use of NSAIDS for the symptomatic relief of medical conditions such as headache or fever is allowed.
* 11. Active infection or unexplained fever > 38.5℃ or last treatment with therapeutic oral or intravenous antibiotics within 2 weeks prior to the first dose of study treatment.

Factors related to the disease

* 12. Known fibrolamellar carcinoma, sarcomatoid HCC or mixed hepatocellular cholangiocarcinoma.
* 13. Has a known active central nervous system (CNS) metastasis.
* 14. Metastatic disease that involves major airways or blood vessels, or centrally located mediastinal tumor masses (<30 mm from the carina) of large volume. Patients with vascular invasion of the portal or hepatic veins may be enrolled.
* 15. Patients with refractory/uncontrolled ascites, pleural effusion or pericardial effusion requiring intervention within 2 weeks before administration of study treatment.
* 16. History of hepatic encephalopathy.
* 17. Liver tumor as a percentage of liver ≥ 50% as judged by the investigator.
* 18. Vp4 type portal vein tumor thrombus and beyond (such as inferior vena cava).
* 19. Untreated or incompletely treated esophageal and/or gastric varices with bleeding or high risk for bleeding or a prior bleeding event due to esophageal and/or gastric varices within 6 months prior to initiation of study treatment.
* 20. Core biopsy or other minor surgical procedure, excluding placement of a vascular access device, within 3 days prior to the first dose of Bevacizumab.
* 21. History of abdominal or tracheoesophageal fistula, gastrointestinal (GI) perforation, or intra-abdominal abscess within 6 months prior to initiation of study treatment.

Diagnostic Assessments

* 22. History of second primary malignancy other than HCC within 5 years prior to screening, except for malignancies with a negligible risk of metastasis or death, such as adequately treated carcinoma in situ of the cervix, non-melanoma skin carcinoma, localized prostate cancer, ductal carcinoma in situ, etc.
* 23. Known allergy or hypersensitivity to any component of the investigational drug product formulation or history of severe allergic anaphylactic reactions to chimeric or humanized antibodies or fusion proteins. Known hypersensitivity to Chinese hamster ovary cell products.
* 24. History of autoimmune disease, including but not limited to myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, vascular thrombosis associated with antiphospholipid syndrome, Wegener's granulomatosis, Sjögren's syndrome, Guillain-Barré syndrome, multiple sclerosis, vasculitis, or glomerulonephritis, etc. Patients with controlled Type 1 diabetes mellitus who are on an insulin regimen are eligible for the study. Patients with a history of autoimmune-related hypothyroidism who are on thyroid-replacement hormone are eligible for the study. Patients with eczema, psoriasis, lichen simplex chronicus, or vitiligo with dermatologic manifestations only (e.g., patients with psoriatic arthritis are excluded) that don't require systemic treatment are eligible for the study. For uncertain autoimmune disease, it could be discussed with the sponsor.
* 25. Prolongation of QTcF (> 470 ms [average of three ECGs], QTc interval corrected by Frederica's formula, QTcF=QT/RR0.33) at screening, and other ECG abnormalities with clinical significance by the judge of the investigator and affect the patient's safety assessment.
* 26. Left ventricle ejection fraction<50%.
* 27. Impaired cardiac function or clinically significant cardiac disease, including but not limit to any one of the following: New York Heart Association class III or IV congestive heart failure, unstable angina, or myocardial infarction within 6 months before administration of the study drug. Any cardiac arrhythmia requiring treatment or intervention. Uncontrolled hypertension (Systolic blood pressure≥150mmHg and/or diastolic blood pressure≥100mmHg).
* 28. Significant vascular disease (e.g., aortic aneurysm requiring surgical repair or recent peripheral arterial thrombosis) within 6 months prior to initiation of study treatment.
* 29. Any serious acute or chronic infection requiring systemic anti-infective therapy (except for viral hepatitis, see exclusion criteria 31-33).
* 30. History of immunodeficiency, including HIV antibody serum test positive, or other acquired/congenital immunodeficiency disease, or active tuberculosis.
* 31. Patients with HBV infection should follow local clinical practice and anti-HBV therapy should be performed to ensure adequate viral suppression. HBV-DNA ≥2000 IU/mL (or equivalent copies/mL) obtained within 14 days prior to initiation of study treatment.
* 32. Patients with HBV and HCV co-infection. If there is only a history of HCV infection, but HCV RNA (-), it is not regarded as HCV infection.
* 33. Patients with active HCV infection (HCV-RNA>103 copies/mL or following local clinical practice) or require concomitant anti-HCV therapy during the study.
* 34. Any other clinically significant comorbidities, such as respiratory, metabolic, congenital, endocrine or central nervous system disease, or any other medical conditions, mental disturbances or social determinants, which in the judgment of the Investigator, could compromise compliance with the protocol, interfere with the interpretation of study results, or predispose the patient to safety risks.

Other Exclusions

* 35. History of allogeneic stem cell transplantation or organ transplantation.
* 36. History of hemoptysis (≥2.5mL of bright red blood per episode) within 1 month prior to initiation of study treatment.
* 37. Evidence of bleeding diathesis or significant coagulopathy (in the absence of therapeutic anticoagulation).
* 38. Current or recent (within 10 days prior to study treatment start) use of aspirin (>325 mg/day) or treatment with dipyramidole, ticlopidine, clopidogrel, and cilostazol.
* 39. Current or recent (within 10 days prior to study treatment start) use of full-dose oral or parenteral anti-coagulants or thrombolytic agents for therapeutic (as opposed to prophylactic) purpose.
* 40. Prophylactic anticoagulation for the patency of venous access devices is allowed provided the activity of the agent results in an INR<1.5×ULN and APTT is within normal limits within 14 days prior to initiation of study treatment.
* 41. For prophylactic use of anti-coagulants or thrombolytic therapies, local label approved dose levels may be used.
* 42. Serious, non-healing or dehiscing wound, active ulcer, or untreated bone fracture.
* 43. Inability to take oral medication or other factors significant preclude adequate absorption of oral medication, such as previously received total gastrectomy, residual gastric dysfunction after subtotal gastrectomy, short bowel syndrome after small bowel resection, active diarrhea or severe irritable bowel syndrome required drug treatment, etc.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Estimated)
Dates: Start 2025-11-14 (Estimated); Primary Completion 2029-03-31 (Estimated); Study Completion 2029-03-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of DLTs | Safety Run-in: At the end of Cycle 1 (each cycle is 21 days)
  Safety Run-in: Incidence of DLTs in Cycle 1
Objective response rate (ORR) | through study completion, an average 21months
  Expansion: Objective response rate (ORR) determined by the investigator according to RECIST v1.1

SECONDARY OUTCOMES:
Progression-Free Survival (PFS) | through study completion, an average 21months
  Progression-Free Survival (PFS) according to RECIST v1.1
Disease control rate (DCR) | through study completion, an average 21months
  Disease control rate (DCR) according to RECIST v1.1
Duration of response (DOR) | through study completion, an average 21months
  Duration of response (DOR) according to RECIST v1.1
Time to progression (TTP) | through study completion, an average 21months
  Time to progression (TTP) :defined as the time from first dose of study drug (Safety Run-in and Expansion) to the first occurrence of imaging assessment of disease progression, as determined by the investigator according to RECIST v1.1
Overall survival (OS) | every 12 weeks from the last dose of treatment for up to 1 year from the subject's last dose of study treatment
  Overall survival (OS): defined as the time from first dose of study drug (Safety Run-in and Expansion) to death from any cause
Incidence and severity of adverse events (AEs), and serious adverse events (SAEs), dose interruption, reduction, or discontinuation of study drug due to toxicity | through study completion, an average 21months
  Incidence and severity of adverse events (AEs), and serious adverse events (SAEs), dose interruption, reduction, or discontinuation of study drug due to toxicity; changes from baseline in physical examinations, Eastern Cooperative Oncology Group (ECOG) performance status (PS), electrocardiograms (ECGs), echocardiograms, laboratory parameters and vital signs.

CONTACTS AND LOCATIONS:
Locations (1):
- Asan Medical Center,, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No